CLINICAL TRIAL: NCT06456957
Title: Fetal Abdominal Subcutaneous Tissue Thickness in Prediction of Fetal Weight in Term Pregnant Women: A Prospective Cohort Study
Brief Title: Fetal Abdominal Subcutaneous Tissue Thickness in Prediction of Fetal Weight in Term Pregnant Women
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Abdallah, Lecturer of Obstetrics and Gynecology, Assiut University
Other Study IDs: FASTT trial
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Ultrasound; Fetal Weight
MeSH Terms: conditions — Fetal Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal Abdominal subcutaneous tissue thickness (FASTT) can be easily measured during the routine ultrasound examination of pregnant women. Numerous reports have shown FASTT measurement to be a good way of evaluating subcutaneous fat tissue.

However, to the best of our knowledge, no studies have investigated the association of FASTT with abnormal fetal growth in nondiabetic. For this reason, in this study we evaluated whether FASTT can predict birth weight or diagnose LGA and/or LBW infants in the third trimester.

DETAILED DESCRIPTION:
The fetal weight assessment by ultrasound is essential in obstetric practice to determine the labor mode, time, and management. It is an important to detect fetal growth abnormalities such as small for gestational age (SGA), fetal growth restriction (FGR) and large for gestational age (LGA) fetuses; thus, it could help in decreasing the perinatal morbidity and mortality rates [1]. Many methods have been introduced to estimate the weight in utero, and many studies have evaluated their effectiveness to detect the most accurate method [2]. Abnormal fetal growth can be diagnosed by ultrasound. Conventional ultrasonic measurements, such as estimated fetal weight (EFW) and abdominal circumference (AC) can distinguish LGA/macrosomia or LBW infants. Many studies have demonstrated that expected fetal weight (EFW) by the traditional techniques is not a reliable indicator of growth abnormalities; consequently several other sono graphic measurements have been proposed [3]. Ultrasound has its limitations despite the use of more than 50 different formulae to estimate fetal weight as their performance is poor at the extremes of fetal weight. There has been emerging interest in studying fetal soft tissue measurements to improve the detection of growth abnormalities [4].

Fetal Abdominal subcutaneous tissue thickness (FASTT) can be easily measured during the routine ultrasound examination of pregnant women. Numerous reports have shown FASTT measurement to be a good way of evaluating subcutaneous fat tissue [5].Furthermore, some researchers have investigated links between FASTT and diabetes [6].

However, to the best of our knowledge, no studies have investigated the association of FASTT with abnormal fetal growth in nondiabetic. For this reason, in this study we evaluated whether FASTT can predict birth weight or diagnose LGA and/or LBW infants in the third trimester.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Gestational age between 37-42 weeks.
3. Accepting to be included in the study

Exclusion Criteria:

1. Pre-gestational diabetes and gestational diabetes.
2. Other medical disorder as hypertensive disorder during pregnancy, cardiac diseases.
3. Congenital fetal malformation affecting birth weight or affecting clavicle.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant women in singleton pregnancy at gestational age between 37 - 40 weeks accepting to be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
sensitivity of measuring Fetal Abdominal Subcutaneous Tissue Thickness | 37-40 weeks gestation
  To evaluate sensitivity of measuring Fetal Abdominal Subcutaneous Tissue Thickness compared to Hadlock formula IV in Prediction of Fetal Weight in Term non-diabetic Pregnant Women in 3rd trimester.

SECONDARY OUTCOMES:
Mode of delivery. | 37-40 weeks gestation
  Vaginal delivery or cesarean section
Gestational age at the time of delivery | 1 week from recruitment
  detection of gestational age at the time of delivery
Neonatal Apgar score | at the time of delivery
  Measure Apgar score for the newborn at 1 minute and 5 minutes
Neonatal birth weight | at the time of delivery
  Measure of Neonatal weight in grams
Neonatal need for NICU | at the time of delivery
  Need for admission of neonate at NICU and Number of days if admitted

REFERENCES:
- [Background] Ebada MA, Elmatboly AM, Baligh G. Intravenous Oxytocin versus Intramuscular Oxytocin for the Management of Postpartum Hemorrhage: A Systematic Review and Meta-Analysis. Curr Drug Res Rev. 2020;12(2):150-157. doi: 10.2174/2589977512666200628013647. PMID 32600245
- [Background] El-Sayed MR, Soliman BS, Zaitoun MM, Shorbaji E, Mohammed RJ. Clinical and ultrasound estimation of fetal weight at term and its accuracy with birth weight. The Egyptian Journal of Hospital Medicine. 2020 Oct 1;81(7):2468-75
- [Background] A Oun Y, M Gebril M, M El-Mazzaly S. Measurement of Fetal Abdominal Subcutaneous Tissue Thickness by Ultrasound in Prediction of Birth Weight at Term Pregnancy. Al-Azhar Medical Journal. 2020 Oct 1;49(4):1653-62.
- [Background] Lu Y, Fu X, Chen F, Wong KKL. Prediction of fetal weight at varying gestational age in the absence of ultrasound examination using ensemble learning. Artif Intell Med. 2020 Jan;102:101748. doi: 10.1016/j.artmed.2019.101748. Epub 2019 Nov 17. PMID 31980089
- [Background] Bethune M, Bell R. Evaluation of the measurement of the fetal fat layer, interventricular septum and abdominal circumference percentile in the prediction of macrosomia in pregnancies affected by gestational diabetes. Ultrasound Obstet Gynecol. 2003 Dec;22(6):586-90. doi: 10.1002/uog.885. PMID 14689530
- [Background] Higgins MF, Russell NM, Mulcahy CH, Coffey M, Foley ME, McAuliffe FM. Fetal anterior abdominal wall thickness in diabetic pregnancy. Eur J Obstet Gynecol Reprod Biol. 2008 Sep;140(1):43-7. doi: 10.1016/j.ejogrb.2008.02.021. Epub 2008 Apr 11. PMID 18406510
- [Background] Lindstrom L, Cnattingius S, Axelsson O, Granfors M. Accuracy and precision of sonographic fetal weight estimation in Sweden. Acta Obstet Gynecol Scand. 2023 Jun;102(6):699-707. doi: 10.1111/aogs.14554. Epub 2023 Mar 25. PMID 36964980
- [Background] Singh, A., Chander, R. and Kumari, S. (2014) Estimation of Fetal Weight and Its Correlation with Actual Birth Weight by Sonographic Measurement of Fetal Abdominal Subcutaneous Tissue Thickness. Journal of Evolution of Medical and Dental Sciences , 3, 9610-9621. https://doi.org/10.14260/jemds/2014/3244